CLINICAL TRIAL: NCT03209947
Title: ULnar Nerve ECHographic Observation (ULNECHO)
Acronym: ULNECHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 29BRC17.0085 ULNECHO
Record Dates: First submitted 2017-07-04; First posted 2017-07-06 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2018-04

CONDITIONS: Ulnar Neuropathies
Keywords: Ulnar Neuropathies; Ultrasound
MeSH Terms: conditions — Ulnar Neuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ulnar nerve ultrasound (Experimental)
  Interventions: Diagnostic Test: Ulnar nerve Ultrasound

INTERVENTIONS:
Diagnostic Test: Ulnar nerve Ultrasound — No drug and no placebo were used in this arm. Patients were followed by Ultrasound approach by measure of ulnar nerve surface

SUMMARY:
There is currently no consensus on the normal ultrasound surface of the ulnar nerve at the elbow. The goal of this study is to study the ulnar nerve surface at the elbow in a population of asymptomatic subjects

DETAILED DESCRIPTION:
100 elbows from 50 patients will be included, from a population of asymptomatic subjects, in order to measure the frequency of ulnar nerve which surface is >8,3 mm².

The measures will be realized centered on the epicondyle : 2 cm higher, and 2 cm lower with 2 echographs (ESAOTE) and 2 observers. An inter and intra observer study will also be realized to determine the reproducibility and reliability of the measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 -to 80 years or older
* Patient without any current or previous pathology on the ulnar nerve
* Patients would be able to consent

Exclusion Criteria:

* Patient under administrative supervision or legal guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Measure of ulnar nerve surface > 8,3 mm ² frequency by Ultrasound | 1 day

SECONDARY OUTCOMES:
Correlation ulnar nerve surface measure of by two doctors | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Letissier H, Dardenne G, Saraux A, Le Nen D, Borotikar B, Jousse-Joulin S. Ultrasound Ulnar Nerve Measurement in a Healthy Population. Rheumatol Ther. 2021 Mar;8(1):457-466. doi: 10.1007/s40744-021-00283-2. Epub 2021 Feb 4. PMID 33543416